CLINICAL TRIAL: NCT03485651
Title: Prospective Collection of Samples for Development of the Natera Ovarian Cancer Detection Assay
Brief Title: Natera Ovarian Cancer Detection Assay
Status: Terminated | Type: Observational
Why Stopped: Poor accrual
Sponsor: Natera, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 15-025-NCT
Record Dates: First submitted 2018-03-09; First posted 2018-04-02 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Adnexal Mass
Keywords: adrexal mass; ovarian cancer; fallopian tube cancer; peritoneal cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples will be retained for research
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to enroll participants who present with an adnexal mass on imaging to develop a non-invasive ovarian cancer assay to distinguish between malignant and benign masses. The study will collect blood, tissue, and health information from these individuals.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to clinic with adnexal mass suspicious of ovarian, fallopian tube, or peritoneal cancer on imaging
* Must be planning surgical resection or biopsy
* Must be treatment naïve
* Must be 18 years or older
* Able to understand and sign a written informed consent document
* Able to provide 40mL of blood (at least 20mL) for each blood draw

Exclusion Criteria:

* Prior removal of either ovary for any reason
* Currently pregnant
* Blood transfusion within 3 months of study enrollment
* History of bone marrow or organ transplant
* Prior history and treatment for any malignancy, with exception of previously treated non-melanoma skin cancer.
* A medical condition that would place subject at risk as a result of the blood donation, including but not limited to bleeding disorders, chronic infectious disease, emphysema or serious anemia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Individuals who present with an adnexal mass on imaging and meet the eligibility criteria. Up to 300 total participants may be enrolled in the study, or until samples from at least 100 malignant cases have been collected.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Compare ctDNA from benign ovarian masses and confirmed ovarian cancers | Up to 60 months or 5 years
  Examine ctDNA between benign ovarian masses and confirmed ovarian cancer cases (based on tumor pathology report). The purpose of this outcome is to determine whether cfDNA could be used to develop a non-invasive ovarian cancer assay to distinguish between malignant and benign masses.

SECONDARY OUTCOMES:
Determine the relationship between quantity of ctDNA and standard prognostic criteria | Up to 60 months or 5 years
  Examine quantity of ctDNA and standard prognostic criteria such as tumor grade, histology and stage of cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Magee-Women's Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No